CLINICAL TRIAL: NCT06088030
Title: Clinical Research on Efficacy and Safety of Arsenic Trioxide Combined With Chemotherapy in p53-mutated Pediatric Cancer Patients：A Prospective，Single-arm, Multi-center Study
Brief Title: Arsenic Trioxide Combined With Chemotherapy for the Treatment of p53-mutated Pediatric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yang Li (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor-Investigator, Yang Li, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYS-202309
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Pediatric Cancer; Li-Fraumeni Syndrome; p53 Mutations
Keywords: Arsenic Trioxide
MeSH Terms: conditions — Neoplasms; Li-Fraumeni Syndrome | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arsenic trioxide combined chemotherapy (Experimental): Patients with p53-mutated pediatric cancer should initially undergo the corresponding first-line chemotherapy regimen. If the patient is evaluated as PD/SD, arsenic trioxide (ATO) will be administered in conjunction with previous conventional chemotherapy on the third day of each treatment cycle.
  Interventions: Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Arsenic trioxide — Patients should be treated with the corresponding first-line chemotherapy regimen first, for example: Neuroblastoma: CAV (cyclophosphamide, pinarubicin, vincristine), PVP (cisplatin, etoposide) ,CT (cyclophosphamide, topotecan).If patients was evaluted as PD/SD after treatments, arsenic trioxide (ATO) will be administered 0.18mg/kg per day over six hours IV daily for ten days in combination with previous chemotherapy regimen on the third day of each treatment cycle. Other pediatric tumors with TP53 mutations not mentioned above will have similar treatment regimens. If the efficacy of the conventional standard chemotherapy regimen is evaluated as PD/SD, then the next course of treatment will be combined with ATO on the basis of the standard chemotherapy regimen.
  Other Names: ATO

SUMMARY:
This prospective, single-arm, multi-center clinical trial aims to explore and evaluate the efficacy and safety of arsenic trioxide combined with chemotherapy for pediatric cancer with p53 mutation.

DETAILED DESCRIPTION:
Germline mutation on tumor suppressor p53 can result in Li-Fraumeni syndrome (LFS), a hereditary condition characterized by the development of multiple cancer types, often at a young or middle age. LFS individuals face a lifetime cancer risk of up to 80-90%, with approximately half of them developing cancer by the age of 30 years. Despite the significantly increased risk of cancer-related morbidity and mortality, clinical management for LFS families is mainly the cancer screenings such as annual whole-body MRIs and the prevention measures such as avoiding exposure to DNA-damaging agents and radiation. Treatment options for LFS patients remain limited. The common LFS treatment regimens involve DNA-damaging chemotherapies and radiotherapies, which often lead to subsequent primary tumors in LFS patients. The susceptibility to second primary tumors is expected since TP53 functions as a haploinsufficient genome guardian. Mutant p53 rescue drugs, which restore tumor-suppressive function to mutant p53 without causing DNA damage, are attractive alternatives, yet no such drugs have been approved for clinical use to date. Unfortunately, the development of LFS-specific treatment drugs has received limited attention from the pharmaceutical industry possibly due to the low prevalence of LFS (occurring in 1 in 5,000 to 1 in 20,000 people worldwide, as evidenced by the lack of clinical trials for LFS treatment.

Different from cancers harboring germline p53 mutation, cancers harboring somatic p53 mutation are being extensively studied in the laboratories and clinics. Somatic p53 mutations can be detected in up to 10 million new cancer incidences per year, making p53 rescue small molecule being one of the most desirable targeted drug in oncology. Many standard treatments (partly) rely on functional wild-type p53 to achieve full treatment efficacy, as supported by the frequently observed higher p53 mutational prevalence in relapsed/refractory cancer patients. Thus, rescue of mutant p53 may (re)sensitize p53-mutant patients to various standard treatments. By 2023, about 25 clinical trials for mutant p53 rescue small molecules, involving over 2000 cancer patients with somatic p53 mutation, are registered on ClinicalTrials.gov.

To date, there have been reports of over twenty generic mutant p53 rescue compounds, with six entering clinical trials, including ATO, APR-246, PAT, COTI-2, PEITC, and Kevetrin. ATO stabilizes the p53 structure by simultaneously binding to the three spatially closed cysteines of the buried ABP pocket, thus strikingly potently stabilizing [16] and rescuing 390 structural p53 mutants, with a preference for the temperature-sensitive (TS) subtype of structural p53 mutants. APR-246 binds to all five exposed cysteines of p53 individually, and the rationale behind stabilizing the p53 structure through the binding of a single exposed cysteine remains inexplicable up to date. PAT shares a similar rescue mechanism to ATO as it also targets the ABP pocket but rescues only the 65 strongest TS p53 mutants due to its weaker stabilization of p53 compared to ATO. The structural rescue mechanisms of COTI-2, PEITC, and Kevetrin are currently unknown. While ATO and PAT are being used to rescue the ATO/PAT-rescuable structural p53 mutations based on their mechanisms and experimental validations, to our knowledge APR-246, COTI-2, PEITC, and Kevetrin are being tested for rescuing all of the p53 mutations in laboratory and clinical settings. However, based on the diversities of the p53 inactivation mechanisms and functional consequences made on p53 mutants, a one-size-fits-all compound that can restore wild-type function to all p53 mutants should not exist. Therefore, p53-rescue treatments in clinical trials is suggested to differentiate p53 mutations and, ideally, experimentally test the rescue effectiveness on the interested mutations before patient treatment.

In this clinical trial, we aim to evaluate the safety and efficacy of ATO in treating cancer patients harboring either germline or somatic p53 mutations. First, we will perform experiments in laboratory to assess the effectiveness of ATO in rescuing the p53 mutations detected in patients. Next, If ATO is effective in rescue a p53 mutation, the patient harboring this mutation (after failures in standard treatments) will be enrolled for clinical trials, using combination treatment of ATO and the standard treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis basis of malignant tumor；
2. Patients not more than 18 years old;
3. Patient has either germline or somatic p53 mutations, which was shown to be partially/completely restored to function by ATO in in vitro experiments (http://www.rescuep53.net);
4. There are measurable lesions;
5. Guardians agreed and signed informed consent.

Exclusion Criteria:

Patients with one or more critical organs failure such as heart, brain, kidney failure.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2031-12-14 (Estimated); Study Completion 2031-12-14 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Four weeks after ATO-combined chemotherapy
  Objective response rate

SECONDARY OUTCOMES:
Progression Free Survival | From the date of patients enrolled to the date of of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Progression Free Survival
Overall survival | From date of randomization to death whichever the cause is, up to 3 years.
  Overall survival
Incidence of Adverse Events | From date of ATO-combined chemotherapy until the date of first documented adverse event, and follow up for 3 years
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yang Li, Professor, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China